CLINICAL TRIAL: NCT02669498
Title: Consequences of Changing Current Standards: Endocrine Status After Routine Fallopian Tube Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 057/12
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Pelvic Surgery; Routine Fallopian Tube Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery with fallopian tube removal (Active Comparator): Patients receiving routine fallopian tube removal during pelvic surgery after randomization.
  Interventions: Procedure: Routine fallopian tube removal
- Surgery without fallopian tube removal (No Intervention): Fallopian tubes are not removed during pelvic surgery after randomization.

INTERVENTIONS:
Procedure: Routine fallopian tube removal — Fallopian tubes are removed by dissection of the Mesosalpinx.
  Arms: Surgery with fallopian tube removal

SUMMARY:
Two recently published articles need to be cited to explain the rationale for our study since both studies conclude with contrary findings: The first one is "The post-reproductive Fallopian tube: better removed?" and the other is termed "Factors associated with age of onset and type of menopause in a cohort of UK women".

In essence, while Dietl et al suggest to remove the Fallopian tube routinely in every hysterectomy and every sterilization procedure after 35 yrs of age, Pokoradi et al showed that pelvic surgical procedures and even simple tubal sterilization are associated with an earlier menopause. Hence, this is an important issue as early menopause leads to adverse health status.

DETAILED DESCRIPTION:
Two study findings lead to conflictive points of view. On the one hand a routine removal of the Fallopian tubes is proclaimed to reduce cancer risk, on the other hand we know that surgical pelvic procedures result in early onset of menopause. Pokoradi et al were not able to distinctively tell which part of pelvic surgery (ie hysterectomy, oophorectomy, salpingectomy, tubal ligation?) is affecting menopause because data was not providing surgical details. Nevertheless, Dietl et al's statement "Timing of menopause and other long-term effects have not been studied yet...thus all negative effects are still speculative"1 can only partly be agreed upon regarding Pokoradi's findings. It might be too early to proclaim a routine Fallopian tube removal as long as there is no data on how much this procedure affects ovarian function. This is further supported by another statement in their study "Although most malignant serous "ovarian" carcinomas originate from the distal Fallopian tube, a smaller proportion of serous cancers as well as endometroid, clear cell, mucinous carcinomas are still thought to arise from ovarian surface epithelium.1" which means the exact impact on cancer prophylaxis can only be estimated due to a lack of studies. Other histopathologic entities might not be influenced by tube removal.

ELIGIBILITY:
Inclusion Criteria:

* benign indication for hysterectomy
* informed consent

Exclusion Criteria:

* Menopause
* Pregnancy
* Previous pelvic surgery (hysterectomy, salpingectomy, tubal ligation,...)
* malignancy
* hormone replacement therapy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-11; Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal changes of FSH pre- and post-operatively | 6 weeks
  Follicle-stimulating hormone (U/l)

SECONDARY OUTCOMES:
Longitudinal changes of AMH | 6 weeks
  AMH (anti-mullerian hormone, U/l)
Longitudinal changes of LH | 6 weeks
  LH (luteinizing hormone, U/l)
Longitudinal changes of E2 | 6 weeks
  E2 (estradiol, U/l)
Longitudinal changes of FSH | 1 year
  Follicle-stimulating hormone (U/l)
Longitudinal changes of AMH | 1 year
  AMH (anti-mullerian hormone, U/l)
Longitudinal changes of LH | 1 year
  LH (luteinizing hormone, U/l)
Longitudinal changes of E2 | 1 year
  E2 (estradiol, U/l)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Mueller, Prof., Study Chair — University Women's Hospital Bern, Switzerland
Locations (2):
- Switzerland (2):
  - Kantonsspital Baden, Baden
  - University Women's Hospital, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dietl J, Wischhusen J, Hausler SF. The post-reproductive Fallopian tube: better removed? Hum Reprod. 2011 Nov;26(11):2918-24. doi: 10.1093/humrep/der274. Epub 2011 Aug 16. PMID 21849300
- [Result] Pokoradi AJ, Iversen L, Hannaford PC. Factors associated with age of onset and type of menopause in a cohort of UK women. Am J Obstet Gynecol. 2011 Jul;205(1):34.e1-13. doi: 10.1016/j.ajog.2011.02.059. Epub 2011 Feb 27. PMID 21514918